CLINICAL TRIAL: NCT04972565
Title: Evaluation and Management of Dyspnea in Hypermobile Ehlers-Danlos Syndrome (hEDS) and Hypermobility Spectrum Disorder (HSD)
Brief Title: Dyspnea in Hypermobile Ehlers-Danlos Syndrome and Hypermobility Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-6346
Record Dates: First submitted 2021-06-25; First posted 2021-07-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hypermobile EDS (hEDS); Hypermobility Syndrome
Keywords: Hypermobile Ehlers Danlos Syndrome; Hypermobility Spectrum Disorder; Dyspnea; Inspiratory Muscle Training; Exercise
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Dyspnea; Motor Activity

STUDY DESIGN:
Intervention Model Description: Hypermobile EDS and HSD participants will be randomized to an inspiratory muscle training group versus usual care. Baseline measures will be compared to 17 age and sex-matched healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care plus Inspiratory Muscle Training (IMT) (Experimental): Participants will attend the standard of care rehabilitation program offered to hEDS and HSD patients at the University Health Network. The program consists of i) an individualized home-based rehabilitation and exercise program (twelve weeks of aerobic, neuromotor, and resistance-based exercises), ii) a self-management education intervention, and iii) a community resource engagement plan. Furthermore, patients attend four on-site sessions (a baseline assessment and three follow-up visits).
  Participants in this group will also be provided with a personalized prescription for an IMT program for eight weeks to be performed in the home environment (two daily IMT sessions of 30 breaths, five days per week). Participants will be virtually supervised by the study team weekly with any adverse events closely monitored. Participants will receive instructions and feedback on how to optimize their home training efforts with direct observation of their IMT practice.
  Interventions: Behavioral: Usual Care plus Inspiratory Muscle Training (IMT)
- Usual Care (No Intervention): Participants will participate in the standard of care rehabilitation program offered to hEDS and HSD patients at the University Health Network.

INTERVENTIONS:
Behavioral: Usual Care plus Inspiratory Muscle Training (IMT) — Participants will receive usual care and will also be provided with a personalized prescription for an IMT program for 8 weeks. Participants will perform two daily IMT sessions of 30 breaths (< 5 minutes/session), 5 days per week in their home environment. IMT intensity will be progressed weekly by 5-10% of the baseline maximal inspiratory pressure if the Borg Dyspnea score is < 7.
  Arms: Usual Care plus Inspiratory Muscle Training (IMT)

SUMMARY:
Individuals with hypermobile Ehlers-Danlos Syndrome (hEDS) and Hypermobility Spectrum Disorders (HSD) often experience dyspnea. Inspiratory Muscle Training (IMT) has been shown to improve dyspnea and respiratory muscle function; however, the impact of IMT in combination with whole-body exercise training on respiratory muscle strength, dyspnea, and daily function remains unknown. The objectives of this research are i) to evaluate dyspnea, respiratory muscle strength and function, ventilatory parameters, and health-related quality of life (HRQL) in individuals with hEDS and HSD compared to healthy age and sex-matched controls, ii) to explore the contributors to dyspnea during exercise with a specific focus on respiratory muscle structure and function in hEDS and HSD patients and healthy controls, and iii) to assess whether the combination of IMT and whole-body exercise training will be more effective than whole-body exercise training alone in improving participant outcomes in hEDS and HSD participants. It is hypothesized that i) hEDS and HSD participants will have lower respiratory muscle strength, higher peripheral airway resistance, lower HRQL, and higher anxiety and depression levels compared to healthy controls, ii) the contributors to increased exercise induced dyspnea will include decreased respiratory muscle strength, increased airway resistance, and greater prefrontal cortical neural activity, and iii) the combination of IMT and whole-body exercise training will be superior to whole-body training alone for improving dyspnea, respiratory muscle strength and endurance, aerobic capacity, HRQL, anxiety, and depression.

DETAILED DESCRIPTION:
Thirty-four hEDS and HSD participants will be recruited from the University Health Network (Toronto, Canada). Participants will have baseline evaluations of dyspnea, pulmonary function tests (i.e., oscillometry, spirometry, and lung volumes), respiratory muscle structure and function (i.e., diaphragm ultrasound and respiratory muscle strength), HRQL, anxiety and depression. Symptom limited cardiopulmonary exercise testing will be utilized to quantify exertional dyspnea using the 10-item Borg dyspnea scale, 18-point qualitative dyspnea assessment scale, peak oxygen uptake (peak VO2), and assessment of dynamic ventilatory parameters. Neural activity in the pre-frontal cortex will be measured during cardiopulmonary exercise testing via functional near-infrared spectroscopy. These baseline measures will be compared to 17 age and sex-matched healthy controls. After baseline assessments, hEDS and HSD participants will be randomized to one of the following groups: i) Usual Care plus IMT: 8 weeks of whole-body exercises (standard care provided to hEDS and HSD patients at the University Health Network) plus a concurrent IMT intervention 5 times per week); ii) Usual Care: 8 weeks of whole-body exercises (as outlined above). After four and eight weeks, participants will have repeat assessments as described below.

Exertional dyspnea is a prevalent and troublesome symptom experienced by individuals living with hEDS and HSD. This study will provide a better understanding of the underlying contributors of dyspnea in hEDS and HSD patients, with a focus on respiratory muscle structure and function, prefrontal cortical neural activity, and ventilatory parameters, both at rest and with exertion.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (≥ 18 years of age)
* New referral to the GoodHope Exercise and Rehabilitation (GEAR) Program at the University Health Network
* Diagnosis of hEDS based on the 2017 diagnostic criteria or diagnosis of HSD (defined as generalized joint hypermobility, chronic pain, and systemic findings to suspect connective tissue underpinnings) with clinical verification by the EDS medical team

Exclusion Criteria:

* Genetic testing confirming the diagnosis of another type of EDS (i.e., vascular EDS, classical EDS)
* Any contraindication to exercise testing (i.e., unstable cardiac disease). Presence of cardiac pacemaker/implantable defibrillator or structural cardiac abnormalities on echocardiogram
* Recent respiratory infection (< 1 month) or known diagnosis of obstructive (i.e., asthma, chronic obstructive pulmonary disease) or restrictive parenchymal lung disease
* History of pneumothorax, otitis media (fluid behind the ear drum), or rupture of tympanic membranes given risk with IMT
* Recent participation in formal exercise training or IMT program (within the last 3 months)
* Persistent symptoms or difficulty tolerating IMT (i.e., breathing difficulties and/or chest pain)
* Diagnosis of severe autonomic dysfunction or postural orthostatic tachycardia syndrome limiting daily physical activity or exercise
* Neuromuscular disease (i.e., myositis, diaphragm paralysis) that may interfere with IMT
* Insufficient English fluency to provide informed consent or ability to follow study protocols
* Self-reported pregnancy
* Inability to connect to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | Change from baseline at 8 weeks
  Maximal inspiratory pressure will be evaluated using standard methods in the pulmonary function laboratory, with the highest value (cm H2O) taken within 10 percent of the other readings as per American Thoracic Society recommendations.

SECONDARY OUTCOMES:
Maximal Expiratory Pressure | Change from baseline at 8 weeks
  Maximal expiratory pressure will be evaluated using standard methods in the pulmonary function laboratory, with the highest value (cm H2O) taken within 10 percent of the other readings as per American Thoracic Society recommendations.
Respiratory Muscle Endurance | Change from baseline at 4 weeks and 8 weeks
  Respiratory muscle endurance (endurance time measured in seconds) will be assessed using a manual threshold loading device (Philips Threshold trainer).
Inspiratory Muscle Training Workload | Through study completion, an average of 8 weeks
  Total IMT workload per session (product of inspiratory muscle force and inhaled volume expressed in Joules) will be extracted from the IMT device in the experimental group.
Inspiratory Muscle Training Load | Through study completion, an average of 8 weeks
  Inspiratory muscle training Load (cm H2O) will be abstracted from the IMT device in the experimental group.
Inspiratory Muscle Training Mean Power | Through study completion, an average of 8 weeks
  Inspiratory muscle training mean power per breath (Watts) will be abstracted from the IMT device in the experimental group.
Inspiratory Muscle Training Mean Volume | Through study completion, an average of 8 weeks
  Inspiratory muscle training mean volume per breath (Litres) will be abstracted from the IMT device in the experimental group.
Medical Research Council Dyspnea Scale | Change from baseline at 8 weeks
  The Medical Research Council Dyspnea Scale will be used to assess the effect of breathlessness on daily activities. The scale comprises five statements that describe the range of respiratory dyspnea from none (Grade 1) to severe with difficulties performing self-care (Grade 5).
Borg Dyspnea Scale | Through study completion, an average of 8 weeks
  The 10-point Borg Dyspnea Scale will be used throughout the study to adjust the intensity of inspiratory muscle training sessions The lowest score (0) corresponds to the sensation of normal breathing (absence of dyspnea) and the highest score (10) corresponds to the maximum possible sensation of dyspnea.
Borg Dyspnea Scale | Change from baseline at 8 weeks
  The 10-point Borg Dyspnea Scale will be used during cardiopulmonary exercise testing to characterize degree of dyspnea. The lowest score (0) corresponds to the sensation of normal breathing (absence of dyspnea) and the highest score (10) corresponds to the maximum possible sensation of dyspnea.
Qualitative Assessment of Dyspnea | Change from baseline at 8 weeks
  The 18-point Qualitative Dyspnea Scale will be ascertained at the end of cardiopulmonary exercise testing. Participants will be presented with a list of 18 descriptors characterizing their dyspnea and will be asked to rank the top three.
Qualitative Assessment of Dyspnea | Change from baseline at 4 weeks and 8 weeks
  The 18-point Qualitative Dyspnea Scale will be ascertained at the end of respiratory muscle endurance testing. Participants will be presented with a list of 18 descriptors characterizing their dyspnea and will be asked to rank the top three.
Oscillometry | Change from baseline at 8 weeks
  Oscillometry will be performed in the pulmonary function laboratory following the protocol from the European Respiratory Society.
Spirometry (Forced Vital Capacity) | Change from baseline at 8 weeks
  Spirometry (forced vital capacity) will be measured in the pulmonary function laboratory following the American Thoracic Society Guidelines.
Spirometry (Forced Expiratory Volume in 1 Second) | Change from baseline at 8 weeks
  Spirometry (forced expiratory volume in 1 second) will be measured in the pulmonary function laboratory following the American Thoracic Society Guidelines.
Lung Volumes (Total Lung Capacity) | Change from baseline at 8 weeks
  Lung volumes (i.e., Total Lung Capacity) will be measured in the pulmonary function laboratory following the American Thoracic Society Guidelines.
Lung Volumes (Inspiratory Capacity) | Change from baseline at 8 weeks
  Lung volumes (i.e., inspiratory capacity) will be measured in the pulmonary function laboratory following the American Thoracic Society Guidelines.
Lung Volumes (Residual Volume) | Change from baseline at 8 weeks
  Lung volumes (i.e., Residual Volume) will be measured in the pulmonary function laboratory following the American Thoracic Society Guidelines.
Diaphragm Thickness | Change from baseline at 8 weeks
  The right hemi-diaphragm thickness will be measured using a 13 megahertz ultrasound transducer.
Diaphragm Thickening Fraction | Change from baseline at 8 weeks
  The right hemi-diaphragm thickening fraction will be measured using a 13 megahertz ultrasound transducer.
Peak Oxygen Uptake During Cardiopulmonary Exercise Testing | Change from baseline at 8 weeks
  Cardiopulmonary exercise test-based assessment of peak oxygen uptake (VO2 peak) will be performed on a cycle ergometer.
Ventilatory Response During Cardiopulmonary Exercise Testing | Change from baseline at 8 weeks
  Ventilatory response will be assessed during cardiopulmonary exercise testing (on a cycle ergometer) with exhaled gas measurements captured breath by breath.
Heart Rate Response During Cardiopulmonary Exercise Testing | Change from baseline at 8 weeks
  Heart rate response will be assessed during cardiopulmonary exercise testing on a cycle ergometer.
Pre-frontal Cortical Neural Activity During Cardiopulmonary Exercise Testing | Change from baseline at 8 weeks
  Oxygenated and total hemoglobin of the prefrontal cortex will be measured with Functional Near Infrared Spectroscopy during cardiopulmonary exercise testing.
Physical Activity Levels | Change from baseline at 4 weeks and 8 weeks
  Physical activity (daily steps) will be measured via a tracking device (Fitbit, San Francisco, USA) for a 7-day period.
Leisure-Time Exercise | Baseline
  Leisure-time exercise will be measured via the 3-item Godin Leisure-Time Exercise Questionnaire - Leisure Score Index. The Leisure Score Index is used to rank individuals from the lowest to highest exercise levels: sedentary (score less than 14 units); moderately active (score of 14-23 units); and active (24 units or more).
Health-Related Quality of Life | Change from baseline at 8 weeks
  The Short-Form 36 Health Survey (SF-36) will be used to assess general health-related quality of life. The SF-36 consists of eight scaled scores (total score ranging from 0 to 100), with lower scores representing lower health-related quality of life.
Depression, Anxiety and Stress Scale | Change from baseline at 8 weeks
  The Depression, Anxiety and Stress Scale (DASS-21) questionnaire has 21 items to assess mood (anxiety, depression, and stress). Each statement for the three domains is given a score of 0 (not applicable) to 3 (applicable most of the time) with scores categorized as follows: Normal, Mild, Moderate, Severe, and Extremely Severe.
Participant Study Recruitment | Over the study period (8 weeks)
  Recruitment-success percentage and reasons for participation/non-participation in the study will be collected.
Participant Retention in the Study | Over the study period (8 weeks)
  Participant retention will be assessed by measuring participant follow-up with testing throughout the study period.
Adherence to Inspiratory Muscle Training Load | Over the intervention period (8 weeks)
  Adherence to the IMT intervention will be tracked electronically via the IMT device (i.e., percentage of the maximal inspiratory pressure prescribed).
Adherence to Inspiratory Muscle Training Days | Over the intervention period (8 weeks)
  Adherence to the IMT intervention will be tracked using a participant log to record the number of training days completed each week.
Adverse Events During Inspiratory Muscle Training Practice (Safety and Tolerability) | Over the intervention period (8 weeks)
  Any adverse events (i.e. prolonged muscle soreness, pneumothorax) with IMT will be assessed throughout the study period.
Participant Satisfaction with the IMT Intervention | Change from baseline at weeks 1, 4 and 8
  A multiple-choice and free-form questionnaire assessing the participants' satisfaction with the IMT intervention will be completed by study participants.

OTHER OUTCOMES:
Electrocardiogram | Baseline
  A 12-Lead Electrocardiogram will be performed in all study participants. The following electrocardiogram parameter (i.e. ST segment) will be assessed to ensure within normal limits before cardiopulmonary exercise testing to ensure no signs of active ischemia.
Chest X-Ray | Baseline
  Chest x-ray will be performed to characterize possible etiologies of dyspnea and exclude any evidence of pneumothorax prior to commencing an IMT program.
Body Mass Index | Change from baseline at 4 weeks and 8 weeks
  Body mass index data (kg/m^2) will be ascertained from clinical records.
Waist Circumference | Change from baseline at 4 weeks and 8 weeks
  Waist circumference (cm) will be ascertained from clinical records.
Demographic Data | Baseline
  A demographic questionnaire will be administered to collect information on age, sex, and ethnicity of the study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Rozenberg, MD, PhD, Principal Investigator — University Health Network/University of Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reychler G, Liistro G, Pierard GE, Hermanns-Le T, Manicourt D. Inspiratory muscle strength training improves lung function in patients with the hypermobile Ehlers-Danlos syndrome: A randomized controlled trial. Am J Med Genet A. 2019 Mar;179(3):356-364. doi: 10.1002/ajmg.a.61016. Epub 2018 Dec 20. PMID 30569502
- [Background] Hakim AJ, Grahame R. Non-musculoskeletal symptoms in joint hypermobility syndrome. Indirect evidence for autonomic dysfunction? Rheumatology (Oxford). 2004 Sep;43(9):1194-5. doi: 10.1093/rheumatology/keh279. No abstract available. PMID 15317957
- [Background] Ayres JG, Pope FM, Reidy JF, Clark TJ. Abnormalities of the lungs and thoracic cage in the Ehlers-Danlos syndrome. Thorax. 1985 Apr;40(4):300-5. doi: 10.1136/thx.40.4.300. PMID 4023980
- [Background] Morgan AW, Pearson SB, Davies S, Gooi HC, Bird HA. Asthma and airways collapse in two heritable disorders of connective tissue. Ann Rheum Dis. 2007 Oct;66(10):1369-73. doi: 10.1136/ard.2006.062224. Epub 2007 Apr 5. PMID 17412739
- [Background] Gazit Y, Nahir AM, Grahame R, Jacob G. Dysautonomia in the joint hypermobility syndrome. Am J Med. 2003 Jul;115(1):33-40. doi: 10.1016/s0002-9343(03)00235-3. PMID 12867232
- [Background] Chatzoudis D, Kelly TJ, Lancaster J, Jones TM. Upper airway obstruction in a patient with Ehlers-Danlos syndrome. Ann R Coll Surg Engl. 2015 Apr;97(3):e50-1. doi: 10.1308/003588414X14055925061793. PMID 26263828
- [Derived] Rozenberg D, Al Kaabi N, Camacho Perez E, Nourouzpour S, Lopez-Hernandez L, McGillis L, Goligher E, Reid WD, Chow CW, Ryan CM, Kumbhare D, Huszti E, Champagne K, Raj S, Mak S, Santa Mina D, Clarke H, Mittal N. Evaluation and Management of Dyspnea in Hypermobile Ehlers-Danlos Syndrome and Generalized Hypermobility Spectrum Disorder: Protocol for a Pilot and Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 20;12:e44832. doi: 10.2196/44832. PMID 36939815